CLINICAL TRIAL: NCT04664868
Title: SphinkeeperTM Procedure for Treating Severe Faecal Incontinence
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christopher Dawoud, Dr.med.univ., Research Fellow, Medical University of Vienna
Other Study IDs: 2338/2019
Record Dates: First submitted 2020-11-30; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Faecal Incontinence
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sphinkeeper™ — Sphinkeeper™ prostheses are self-expandable solid prostheses, made of inert Hyexpan (polyacrylonitrile) and are inserted into the intersphincteric anal groove.

SUMMARY:
Patients, aged 18 - 90 years, undergoing sphinkeeper operation at the Department of General Surgery at the Medical University of Vienna are enrolled into our study. Primary endpoints is the functional outcome as well as movement, migration and extrusion of sphinkeeper prostheses after implantation by endoluminal ultrasound and manometrical examination.

DETAILED DESCRIPTION:
The Sphinkeeper™ implantation for fecal incontinence is a novel surgical procedure with limited data on its clinical efficacy. Therefore, we aimed to assess the functional outcome following Sphinkeeper™ surgery in patients with refractory FI.

Patients with FI, who met the inclusion criteria were enrolled to our study and received Sphinkeeper™ implantation. Functional outcome and quality of life was evaluated by standard questionnaires before and after surgery. In the routine check-up patients received endoanal ultrasound and anorectal manometry.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 90 years, undergoing sphinkeeper operation at the Department of General Surgery, Medical University of Vienna
* Ability and willingness to understand and comply with study interventions and restrictions.
* Voluntarily signed informed consent after full explanation of the study to the participant.

Exclusion Criteria:

* Any physical or mental disorder, which could interfere with the participant's safety during the clinical trial or with the study objectives
* Inability to communicate well with the investigator due to language problems or reduced mental development
* Inability or unwillingness to give written informed consent

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Candidates for sphinkeeper operations due to fecal incontinence will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Faecal incontinence assessment | six months
  Episodes and number of faecal incomtinence and stool form with faecal incontinence were assessed using the Vaizey incontinence score (range 0-22, higher numbers mean severe incontinence forms)

SECONDARY OUTCOMES:
Psychological und physical well-being | six months
  The Psychological und physical well-being before and after implantation of Sphinkeeper was assessed using the SF12 standardized questionnaire (range 0-100; higher scores= Better quality of life)
Migration of Sphinkeeper prostheses | six months
  The Migration of Sphinkeeper prostheses were analyzed using endoanal ultrasound one and six months after implantation. The prostheses will be categorized by their position in relation to the anal canal axis. (Grade of rotation to the anal canal axis)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Riss, Prof.MD, Study Chair — Medical University of Vienna, Head of Pelvic Floor surgery
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
IPD can be shared just in anonymised form in case of an ethical agreement with other researchers.